CLINICAL TRIAL: NCT01246791
Title: A Single Dose Pharmacokinetics Study of NPC-01 (1mg Norethisterone and 0.02mg Ethynyl Estradiol) in Healthy Female Volunteers
Brief Title: Pharmacokinetics of NPC-01 After Single Oral Administration in Healthy Female Volunteers
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Nobelpharma (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NPC-01-3
Record Dates: First submitted 2010-11-18; First posted 2010-11-23 (Estimated); Results first posted 2014-06-17 (Estimated); Last update posted 2025-06-17 (Actual); Status verified 2025-06

CONDITIONS: Healthy
Keywords: NPC-01; Pharmacokinetics; Healthy female volunteer; Norethisterone; Ethinyl Estradiol
MeSH Terms: interventions — Norethindrone; Ethinyl Estradiol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- NPC-01 (Experimental): Single oral administration of NPC-01
  Interventions: Drug: NPC-01

INTERVENTIONS:
Drug: NPC-01 — NPC-01, contains 1mg norethisterone and 0.02mg ethinyl estradiol will be administered orally under the fasting condition
  Other Names: Norethisterone and Ethinyl Estradiol

SUMMARY:
The purpose of this study is to assess the pharmacokinetic profiles of norethisterone and ethinyl estradiol after single oral administration of NPC-01 in healthy female volunteers.

Pharmacokinetics of norethisterone and ethinyl estradiol will be evaluated on the basis of AUC, Cmax, tmax, t1/2, MRT, kel and AUC∞.

ELIGIBILITY:
Inclusion Criteria:

* Healthy female aged between 20 to 35 years
* BMI:18.0-26.0

Exclusion Criteria:

* Females who are pregnant
* Drug use affecting sex hormone secretion

Ages: 20 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2010-11; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Takefumi Matuo, MD, Principal Investigator — Hyogo Prefectural AWAJI Hospital

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Thirty healthy female are screened for this study. Appropriate subjects who satisfy inclusion criteria were enrolled for this study.
Period: Overall Study
Arm/Group | NPC-01
Started | 12
Completed | 12
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | NPC-01
Number analyzed (Participants) | 12
Age, Continuous [Mean (Standard Deviation); unit: years] | 27.3 (5.0)
Sex/Gender, Customized [Number; unit: participants]
  Female | 12
Height [Mean (Standard Deviation); unit: cm] | 158.98 (6.31)
Body weight [Mean (Standard Deviation); unit: kg] | 54.46 (9.70)

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Plasma Concentration Versus Time Curve (AUC) on Norethisterone of NPC-01
Description: Multiple blood samples will obtains at pretreatment(0 hour), 0.5, 1.0, 1.5, 2.0, 4.0, 6.0, 9.0, 12.0 and 24.0 hours after dosing of NPC-01(1mg norethisterone and 0.02mg ethinyl estradiol) and determination of area under the plasma concentration versus time curve (AUC) of norethisterone that are active substances of NPC-01.
Time Frame: 0, 0.5, 1.0, 1.5, 2.0, 4.0, 6.0, 9.0, 12.0, 24.0 hours after single dosing of NPC-01
Measure: Mean (Standard Deviation); unit: ng･hr/mL
Arm/Group | NPC-01
Number analyzed (Participants) | 12
ng･hr/mL | 69.183 (36.316)

2. Primary Outcome: Area Under the Plasma Concentration Versus Time Curve (AUC) on Ethinyl Estradiol of NPC-01
Description: Multiple blood samples will obtains at pretreatment(0 hour), 0.5, 1.0, 1.5, 2.0, 4.0, 6.0, 9.0, 12.0 and 24.0 hours after dosing of NPC-01(1mg norethisterone and 0.02mg ethinyl estradiol) and determination of area under the plasma concentration versus time curve (AUC) of ethinyl estradiol that are active substances of NPC-01.
Time Frame: 0, 0.5, 1.0, 1.5, 2.0, 4.0, 6.0, 9.0, 12.0, 24.0 hours after single dosing of NPC-01
Measure: Mean (Standard Deviation); unit: pg･hr/mL
Arm/Group | NPC-01
Number analyzed (Participants) | 12
pg･hr/mL | 368.123 (170.882)

3. Primary Outcome: Peak Plasma Concentration (Cmax) on Norethisterone of NPC-01
Description: Multiple blood samples will obtains at pretreatment(0 hour), 0.5, 1.0, 1.5, 2.0, 4.0, 6.0, 9.0, 12.0 and 24.0 hours after dosing of NPC-01(1mg norethisterone and 0.02mg ethinyl estradiol) and determination of peak plasma concentration (Cmax) of norethisterone that are active substances of NPC-01.
Time Frame: 0, 0.5, 1.0, 1.5, 2.0, 4.0, 6.0, 9.0, 12.0, 24.0 hours after single dosing of NPC-01
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | NPC-01
Number analyzed (Participants) | 12
ng/mL | 12.481 (6.205)

4. Primary Outcome: Peak Plasma Concentration (Cmax) on Ethinyl Estradiol of NPC-01
Description: Multiple blood samples will obtains at pretreatment(0 hour), 0.5, 1.0, 1.5, 2.0, 4.0, 6.0, 9.0, 12.0 and 24.0 hours after dosing of NPC-01(1mg norethisterone and 0.02mg ethinyl estradiol) and determination of peak plasma concentration (Cmax) of ethinyl estradiol that are active substances of NPC-01.
Time Frame: 0, 0.5, 1.0, 1.5, 2.0, 4.0, 6.0, 9.0, 12.0, 24.0 hours after single dosing of NPC-01
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | NPC-01
Number analyzed (Participants) | 12
pg/mL | 55.783 (17.201)

5. Primary Outcome: Time to Peak Plasma Concentration (Tmax) on Norethisterone of NPC-01
Description: Multiple blood samples will obtains at pretreatment(0 hour), 0.5, 1.0, 1.5, 2.0, 4.0, 6.0, 9.0, 12.0 and 24.0 hours after dosing of NPC-01(1mg norethisterone and 0.02mg ethinyl estradiol) and determination of time to peak plasma concentration (Tmax) of norethisterone that are active substances of NPC-01.
Time Frame: 0, 0.5, 1.0, 1.5, 2.0, 4.0, 6.0, 9.0, 12.0, 24.0 hours after single dosing of NPC-01
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | NPC-01
Number analyzed (Participants) | 12
hours | 1.81 (0.79)

6. Primary Outcome: Time to Peak Plasma Concentration (Tmax) on Ethinyl Estradiol of NPC-01
Description: Multiple blood samples will obtains at pretreatment(0 hour), 0.5, 1.0, 1.5, 2.0, 4.0, 6.0, 9.0, 12.0 and 24.0 hours after dosing of NPC-01(1mg norethisterone and 0.02mg ethinyl estradiol) and determination of time to peak plasma concentration (Tmax) of ethinyl estradiol that are active substances of NPC-01.
Time Frame: 0, 0.5, 1.0, 1.5, 2.0, 4.0, 6.0, 9.0, 12.0, 24.0 hours after single dosing of NPC-01
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | NPC-01
Number analyzed (Participants) | 12
hours | 1.50 (0.43)

7. Primary Outcome: Plasma Half Life (t1/2) on Norethisterone of NPC-01
Description: Multiple blood samples will obtains at pretreatment(0 hour), 0.5, 1.0, 1.5, 2.0, 4.0, 6.0, 9.0, 12.0 and 24.0 hours after dosing of NPC-01(1mg norethisterone and 0.02mg ethinyl estradiol) and determination of plasma Half life (t1/2) of norethisterone that are active substances of NPC-01.
Time Frame: 0, 0.5, 1.0, 1.5, 2.0, 4.0, 6.0, 9.0, 12.0, 24.0 hours after single dosing of NPC-01
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | NPC-01
Number analyzed (Participants) | 12
hours | 7.357 (1.863)

8. Primary Outcome: Plasma Half Life (t1/2) on Ethinyl Estradiol of NPC-01
Description: Multiple blood samples will obtains at pretreatment(0 hour), 0.5, 1.0, 1.5, 2.0, 4.0, 6.0, 9.0, 12.0 and 24.0 hours after dosing of NPC-01(1mg norethisterone and 0.02mg ethinyl estradiol) and determination of plasma Half life (t1/2) of ethinyl estradiol that are active substances of NPC-01.
Time Frame: 0, 0.5, 1.0, 1.5, 2.0, 4.0, 6.0, 9.0, 12.0, 24.0 hours after single dosing of NPC-01
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | NPC-01
Number analyzed (Participants) | 12
hours | 5.499 (2.207)

9. Primary Outcome: Mean Residence Time (MRT) on Norethisterone of NPC-01
Description: Multiple blood samples will obtains at pretreatment(0 hour), 0.5, 1.0, 1.5, 2.0, 4.0, 6.0, 9.0, 12.0 and 24.0 hours after dosing of NPC-01(1mg norethisterone and 0.02mg ethinyl estradiol) and determination of mean residence time (MRT) of norethisterone that are active substances of NPC-01.
Time Frame: 0, 0.5, 1.0, 1.5, 2.0, 4.0, 6.0, 9.0, 12.0, 24.0 hours after single dosing of NPC-01
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | NPC-01
Number analyzed (Participants) | 12
hours | 6.340 (0.459)

10. Primary Outcome: Mean Residence Time (MRT) on Ethinyl Estradiol of NPC-01
Description: Multiple blood samples will obtains at pretreatment(0 hour), 0.5, 1.0, 1.5, 2.0, 4.0, 6.0, 9.0, 12.0 and 24.0 hours after dosing of NPC-01(1mg norethisterone and 0.02mg ethinyl estradiol) and determination of mean residence time (MRT) of ethinyl estradiol that are active substances of NPC-01.
Time Frame: 0, 0.5, 1.0, 1.5, 2.0, 4.0, 6.0, 9.0, 12.0, 24.0 hours after single dosing of NPC-01
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | NPC-01
Number analyzed (Participants) | 12
hours | 5.161 (1.504)

11. Primary Outcome: Elimination Rate Constant (Kel) on Norethisterone of NPC-01
Description: Multiple blood samples will obtains at pretreatment(0 hour), 0.5, 1.0, 1.5, 2.0, 4.0, 6.0, 9.0, 12.0 and 24.0 hours after dosing of NPC-01(1mg norethisterone and 0.02mg ethinyl estradiol) and determination of elimination rate constant (kel) of norethisterone that are active substances of NPC-01.
Time Frame: 0, 0.5, 1.0, 1.5, 2.0, 4.0, 6.0, 9.0, 12.0, 24.0 hours after single dosing of NPC-01
Measure: Mean (Standard Deviation); unit: hr^-1
Arm/Group | NPC-01
Number analyzed (Participants) | 12
hr^-1 | 0.101 (0.029)

12. Primary Outcome: Elimination Rate Constant (Kel) on Ethinyl Estradiol of NPC-01
Description: Multiple blood samples will obtains at pretreatment(0 hour), 0.5, 1.0, 1.5, 2.0, 4.0, 6.0, 9.0, 12.0 and 24.0 hours after dosing of NPC-01(1mg norethisterone and 0.02mg ethinyl estradiol) and determination of elimination rate constant (kel) of ethinyl estradiol that are active substances of NPC-01.
Time Frame: 0, 0.5, 1.0, 1.5, 2.0, 4.0, 6.0, 9.0, 12.0, 24.0 hours after single dosing of NPC-01
Measure: Mean (Standard Deviation); unit: hr^-1
Arm/Group | NPC-01
Number analyzed (Participants) | 12
hr^-1 | 0.141 (0.043)

ADVERSE EVENTS:
Time Frame: From initiation of study drug administration to follow up visit (day 7±1 day)
Arm/Group | NPC-01
Serious Adverse Events (participants affected / at risk) | 0/12
Other Adverse Events (participants affected / at risk) | 3/12
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | NPC-01 (N=12)
Headache (Nervous system disorders) | 1 (1)
Metrorrhagia (Reproductive system and breast disorders) | 2 (2)
Blood iron decreased (Investigations) | 1 (1)
White blood cell count decreased (Investigations) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
There is an agreement between the sponsor and PI that no restricts the PI's right but need to discuss the timing of publish date of trial results after the trial is completed.